CLINICAL TRIAL: NCT02671292
Title: Preventing Obesity in Military Communities-Adolescents
Acronym: POMC-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MPS-72-3248; R01DK104115 (NIH)
Record Dates: First submitted 2015-07-09; First posted 2016-02-02 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Overweight; Binge Eating
Keywords: Loss of Control Eating; Binge Eating; Obesity; Prevention; Interpersonal Psychotherapy; Adolescent
MeSH Terms: conditions — Obesity; Overweight; Bulimia | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpersonal Psychotherapy (IPT-WG) (Experimental): IPT-WG targets the difficult social functioning and stressful events that are associated with loss of control eating and that are highly relevant to the adolescent children of military personnel.
  Interventions: Behavioral: Interpersonal Psychotherapy
- Health Education (HE) (Active Comparator): HE improves knowledge on various health topics including, alcohol, drug and tobacco use, depression and suicide, nutrition and body image, nonviolent conflict resolution, sun safety, exercise, and domestic violence.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — IPT-WG involves one initial 1.5-hour individual session, and 12 weekly 90-minute group sessions. The IPT-WG group sessions follow 3 phases (initial, middle, and termination) and use the interpersonal inventory to identify interpersonal problems that might be contributing to or exacerbated by LOC eating. A framework of common problem areas is used to teach interpersonal problem-solving and communication skills and educate youth about risk factors for excessive weight gain and warning signs such as eating in response to negative affect as opposed to hunger, or feeling a sense of LOC while eating.
  Arms: Interpersonal Psychotherapy (IPT-WG)
Other: Health Education — The HE group is based upon the "HEY-Durham" health program designed by researchers at Duke University. This program, designed to be delivered to youth attending community high schools, was adapted to a 12-week program (each session is 90 minutes). Additionally, individuals will attend a pre-group individual meeting with the group leaders to review family health history.The curriculum includes focus on various health topics, including alcohol, drug and tobacco use, depression and suicide, nutrition and body image, nonviolent conflict resolution, sun safety, exercise, and domestic violence. Session content will be largely identical for boys and girls, with the exception of gender-specific videos and articles (e.g., on body image), which will be tailored for each sex.
  Arms: Health Education (HE)

SUMMARY:
To determine whether reducing loss of control eating (LOC) with Interpersonal Psychotherapy-Weight Gain (IPT-WG) will be effective for adolescent military-dependents who report such behavior. The investigators will examine whether IPT-WG influences body weight gain trajectories and prevents worsening disordered eating, psychosocial problems, and metabolic functioning among military dependents at heightened risk for adult obesity and disordered eating. This study will provide key efficacy data for a new promising obesity prevention program for youth from military families.

DETAILED DESCRIPTION:
The prevalence of overweight among military personnel and their dependents is at a rate similar to that of the civilian population. Nearly 30% of adolescent dependents are overweight, including approximately 15-17% who are obese, placing them at high risk for impairments in metabolic functioning, type 2 diabetes, and adult obesity. Youth who are overweight (body mass index, kg/m2, BMI ≥ 85th percentile) are at high risk for excess weight gain as they grow. Since effective weight loss and maintenance treatments are rare, prevention may be the most important approach to reducing the high prevalence of obesity. To date, most pediatric obesity prevention programs have been met with limited success. To address those at greatest risk for obesity, more targeted approaches may be required. There is a need to reduce prospectively identified risk factors in order to prevent excess weight gain in youth at high risk for adult obesity. The most common disordered eating behavior among overweight adolescents is loss of control (LOC) eating, during which the feeling of being unable to stop eating is experienced. LOC eating predisposes youth to gain excessive weight and fat. Thus, LOC eating is likely to be an important contributor to obesity in susceptible individuals. Decreasing LOC in adolescents may prevent excess weight gain. Investigators at the Uniformed Services University of the Health Sciences (USUHS) is in partnership with Ft. Belvoir Community Hospital (FBCH) and Walter Reed National Military Medical Center (WRNMMC) to test the effectiveness of IPT-WG to slow the trajectory of weight gain in overweight adolescent boys and girls who report LOC and prevent worsening disordered eating and metabolic functioning. The unique stress burdening the children of military personnel while the country is at war suggests that obesity prevention programs targeting interpersonal stress and promoting positive social functioning may be especially timely in this population. It is hypothesized that IPT-WG will decrease LOC eating and related eating behaviors and, in turn, prevent excess weight gain and the development of exacerbated disordered eating in adolescent children of military personnel. Secondary to the prevention of excess weight gain, youth will experience improvements in metabolic functioning.

ELIGIBILITY:
Adolescent Inclusion Criteria:

1. Age between 12 and 17 years (at the start of the study)
2. BMI at or above the 85th percentile for age and sex
3. English-speaking
4. Ability to complete study procedures, including the ability to participate in a group
5. > 1 episode of LOC eating during the 3 months prior to assessment
6. Must have a parent(s) enrolled in TRICARE at the time of study initiation

Parent Inclusion Criteria:

1.The consenting parent or caregiver must be able to comprehend English.

Adolescent Exclusion Criteria:

1. Presence of a chronic major medical illness: renal, hepatic, gastrointestinal, endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication).
2. Presence of a documented, obesity-related medical complication that would require a more aggressive weight loss intervention approach: type 2 diabetes, hyperlipidemia, hypertension, fasting hyperglycemia, or nonalcoholic steatohepatitis.
3. Self-reported current pregnancy, current breast-feeding, or recently pregnant girls (within 1 year of delivery).
4. Current, regular use of prescription medications that affect appetite, mood, or body weight: currently prescribed SSRI's, neuroleptics, tricyclics, stimulants, or any other medication known to affect appetite, mood, or body weight. For girls, oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting the prevention groups. Medication use for non-serious conditions (e.g., acne) will be considered on a case-by-case basis.
5. Current involvement in psychotherapy or a structured weight loss program.
6. Weight loss during the past two months for any reason exceeding 3% of body weight.
7. Current anorexia nervosa or bulimia nervosa as determined by documented medical history or if uncovered during K-SADS semi-structured interview. Current binge eating disorder (BED) will be permitted, although adolescents will be informed that they have an eating disorder and have the option to participate in the study or seek outside treatment (and not participate in the study).
8. Individuals who have major depressive disorder, psychoses, current substance or alcohol abuse, conduct disorder, as determined by Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) semi-structured interview and as defined by criteria outlined in the DSM-5, or any other DSM psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.

Parent Exclusion Criteria:

1. None

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Participant Weight | Change in weight from baseline to 3 years post-treatment
  Weight will be measured

SECONDARY OUTCOMES:
Presence of binge eating | Change in presence of binge eating from baseline to 1 year post-treatment
  The Eating Disorder Examination (EDE) will be administered to assess for the presence of binge eating. The EDE identifies three types of eating episodes: objective binge eating (overeating with LOC), subjective binge eating (LOC without objective overeating as assessed by the interviewer, but viewed as excessive by the interviewee), and objective overeating (overeating without LOC), as well as the range of compensatory behaviors described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
Waist Circumference | Change in waist circumference from baseline to 3 years post-treatment
  Waist circumference will be measured using a flexible measuring tape.
Blood Pressure | Change in blood pressure from baseline to 3 years post-treatment
  Blood pressure will be measured using an automatic blood pressure cuff.
Triglycerides | Change in triglycerides from baseline to 3 years post-treatment
  Blood will be drawn to collect a sample for the measurement of triglycerides.
HDL Cholesterol | Change in HDL cholesterol from baseline to 3 years post-treatment
  Blood will be drawn to collect a sample for the measurement of HDL.
Insulin Function | Change in insulin sensitivity from baseline to 3 years post-treatment
  Blood will be drawn to collect a sample for the measurement of insulin.
Glucose | Change in glucose from baseline to 3 years post-treatment
  Blood will be drawn to collect a sample for the measurement of glucose.
Hemoglobin A1c | Change in hemoglobin A1c from baseline to 3 years post-treatment
  Blood will be drawn to collect a sample for the measurement of hemoglobin A1c.
BMI Percentile | Change in BMI percentile from baseline to 3 years post-treatment
  Height and weight will be measured and BMI percentile calculated

CONTACTS AND LOCATIONS:
Overall Officials: Marian Tanofsky-Kraff, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solomon S, Shank LM, Lavender JM, Neyland MKH, Gallager-Teske J, Markos B, Haynes H, Repke H, Rice AJ, Sbrocco T, Wilfley DE, Schvey NA, Jorgensen S, Ford B, Ford CB, Haigney M, Klein DA, Quinlan J, Tanofsky-Kraff M. The Relationship Between Anxiety, Coping, and Disordered-Eating Attitudes in Adolescent Military-Dependents at High-Risk for Excess Weight Gain. Mil Psychol. 2023;35(2):95-106. doi: 10.1080/08995605.2022.2083448. Epub 2022 Jun 21. PMID 36968637

DOCUMENTS (1):
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT02671292/ICF_000.pdf